CLINICAL TRIAL: NCT06614855
Title: A Phase IB 2 Dose Trial of IRS-1 HSV C134 (IND 17296) Administered Intratumorally in Patients With Recurrent Malignant Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: James Markert, MD (Other)
Responsible Party: Sponsor-Investigator, James Markert, MD, Chair, Department of Neurosurgery, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013560; HT94252310805 (Other: DoD)
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Glioblastoma (GBM); Astrocytoma; Astrocytoma, Grade III; Astrocytoma, Grade IV; Gliosarcoma, Adult; Gliosarcoma of Brain
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Initial Treatment (Experimental): Patients will undergo a contrasted MRI scan to determine the site for stereotactic biopsy. For dose #1, patients will be treated under monitored local anesthesia, or at the surgeon's discretion, under general anesthesia. Patients will then undergo stereotactic biopsy of their tumor. While evidence of radiation damage or necrosis may be present on the frozen section, inoculation with C134 will only proceed if viable, recurrent glioma is also present on the frozen section. The dose level of C134 will be 1 x 105 plaque forming units (pfu). Virus will be inoculated via catheters placed stereotactically in enhancing regions of tumor or immediately adjacent in non-enhancing tumor infiltrated regions at up to 5 different loci (each injection over 2 minutes). Catheters will be removed directly after administration for treatment 1.
  Interventions: Drug: C134
- 2nd Treatment (Experimental): Before dose #2 administration, patients will undergo preoperative assessment of their disease status.
  If they are deemed to have had a complete response (CR), no treatment will be undertaken until there is evidence of a possible recurrence. If this does not occur until after week 16, the patient's situation will be discussed with the DSMB and a decision made about possible second treatment.
  If the patient has had a partial response or stable disease, and their tumor remains less than 5.5 cm in size, they wil lbe treated with stereotactic biopsy using the same technique described for dose #1
  If the patient has suffered progression or peudoprogression, or if in the estimation of the surgeon it is not safe to perform inoculation alone, they will undergo craniotomy for resection of the tumor.
  Interventions: Drug: C134

INTERVENTIONS:
Drug: C134 — Initial Treatment . C134 Dose #1
  Arms: Initial Treatment
Drug: C134 — 2nd Treatment. C134 Dose #2
  Arms: 2nd Treatment

SUMMARY:
The purpose of this study is to determine how safe and how well-tolerated the experimental study drug, C134 is when administered twice into the brain where the tumor is located. This is a Phase IB 2 dosing study. All the patients who take part in this study will receive the same type of experimental treatment. There is no "placebo" in this study. The patient will receive the dose of C134 administered, which will be added in the tumor infiltrated tissue in the area of the resection cavity. Anywhere from 4-12 patients are expected to take part in the study; the final number will depend on the safety results.

DETAILED DESCRIPTION:
This study is divided into the following sections, also called phases: the Initial Screening Phase, Initial Treatment Phase, Initial Treatment Follow-up Phase, 2nd Treatment Screening Phase, 2nd Treatment Phase, 2nd Treatment Follow-up Phase. Before the subject can participate in the study, tests will be performed to make sure that the subject qualifies for the study. This is called the Initial Screening Phase. If the subject qualifies for the study they will then enter the Initial Treatment Phase which is the phase where they will receive the study drug and then enter the Initial Follow-up Phase. If there are signs of progression, the subject will be entered into the 2nd Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed recurrent/progressive glioblastoma multiforme, Grade 3 or Grade 4 astrocytoma, or gliosarcoma.
* Prior therapy. Patients must have failed a course of external beam radiotherapy to the brain at least 4 weeks prior to enrollment.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of C134 in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* Karnofsky Performance Status ≥70%.
* Life expectancy of greater than 4 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/ μl
  * absolute neutrophil count ≥ 1,500/ μl
  * platelets ≥ 100,000/ μl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Residual lesion must be ≥1.0 cm in diameter as determined by MRI.
* The effects of C134 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the first six months after receiving C134. Because it is currently unknown if C134 can be transmitted by sexual contact, a barrier method of birth control should be employed. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Females of childbearing potential must not be pregnant; this will be confirmed by a negative serum pregnancy test within 14 days prior to starting study treatment.
* Steroid use is allowed as long as dose has not increased within 2 weeks of scheduled initial C134 administration. Whenever possible, the patient should be on a steroid dose that is equivalent to a dexamethasone dose of ≤ 2mg daily at study entry and initial treatment.

Exclusion Criteria:

* Patients who have had chemotherapy, cytotoxic therapy, immunotherapy or gene therapy within 6 weeks prior to entering the study, surgical resection within 4 weeks prior to entering the study, or have received experimental viral therapy at any time (e.g., adenovirus, retrovirus or herpesvirus* protocol unless approved by DSMB). Also, those who have not recovered from adverse events due to therapeutic interventions administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents (except C134 per protocol).
* Enhancing tumor diameter larger than 5.5 cm for initial treatment or subsequent treatment if only stereotactic biopsy is planned. If resection is planned at the time of second treatment, there is no limit to tumor size at that time. In other words, if the tumor enlarges from less than 5.5 cm to larger than 5.5 cm during the interval between treatment one and two, as long as a resection is planned along with treatment two, no limit in size is present (Note: this size limitation has been derived from experience with prior oHSV therapeutics in malignant glioma).
* History of allergic reactions or CTCAE version 5.0 Grade IV toxicity attributed to C134 or compounds of similar biologic composition to C134.
* Tumor involvement which would require ventricular, brainstem, basal ganglia, occipital lobe, or posterior fossa inoculation or would require access through a ventricle in order to deliver treatment. Additionally, patients with bilateral enhancing tumor are not eligible.
* Prior history of encephalitis, multiple sclerosis. Patient with other active CNS infections are also excluded.
* Active oral herpes lesion.
* Concurrent therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery. Also, psychiatric illness/social situations that would limit compliance with study requirements.
* Required steroid increase within 2 weeks of initial scheduled C134 administration. When possible, the patient should be on a dexamethasone equivalent dose of ≤ 2mg daily at the time of treatment.
* Known history of allergic reaction to IV contrast material that is not amenable to pre-treatment by UAB protocol.
* Have a pacemaker, ferro-magnetic aneurysm clips, metal infusion pumps, metal or shrapnel fragments, or certain types of stents that preclude MRI.
* Received Bevacizumab (Avastin) therapy within 4 weeks of scheduled C134 administration.

Excluded patient groups:

* Pregnant women are excluded from this study because C134 is a viral oncolytic therapy with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with C134 breastfeeding should be discontinued if the mother is treated with C134.
* Immune deficient, because patients with immune deficiency will be unable to mount the anticipated immune response underlying this therapeutic rationale, HIV-seropositive patients are excluded from this study. Other treatment studies for this disease that are less dependent on the patients' immune response are more appropriate for HIV-seropositive patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety of a two dose intracerebral injection of C134 virus | Enrollment - 12 Month
  Adverse events will be monitored and any changes in status will be recorded for each patient as outlined in CTCAE v4.0 reporting requirements.

SECONDARY OUTCOMES:
Time to survival | Enrollment - 12 Month
  Patients survival will be recorded (Kaplan-Meier)
Time to progression | Enrollment - 12 Month
  Patients will receive contrast-enhanced MRI to monitor progression (changes in tumor volume or tumor enhancement assessed by the iRANO criteria). As indicated in the criteria, biopsy and/or resection may be performed in instances of uncertainty. Determination of time to progression (in months) will be recorded for each patient and median progression-free survival will be calculated for the entire cohort (Kaplan-Meier).
Composition of the white blood cells | Enrollment - 12 Month
  White blood cell subset analysis by FACS, as a percent of total white blood cell number.
Measurement of HSV Titer | Enrollment - 12 Month
  Detection and quantification of HSV antibody titer via ELISA, pfu/mL.
Measure interferon levels | Enrollment - 12 Month
  Intracellular lymphocyte interferon levels will be assessed by FACS analysis ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No